CLINICAL TRIAL: NCT02416271
Title: Teriparatide Compared With Alendronate on Spine Bone Mineral Density in Postmenopausal Women With Osteoporosis
Brief Title: The Forteo Alendronate Comparator Trial
Acronym: FACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4943; B3D-MC-GHBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Alendronate; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teriparatide (Experimental): 20 micrograms per day teriparatide subcutaneous (SC) injection plus oral placebo for 18 months.
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: Placebo-Oral
- Alendronate (Active Comparator): 10 milligrams/day alendronate orally plus SC injection placebo for 18 months.
  Interventions: Drug: Alendronate; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: Placebo-SC

INTERVENTIONS:
Drug: Teriparatide — Administered SC
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: Alendronate — Administered orally
  Arms: Alendronate
Dietary Supplement: Calcium — Administered orally
Dietary Supplement: Vitamin D — Administered orally
Drug: Placebo-Oral — Administered orally
  Arms: Teriparatide
Drug: Placebo-SC — Administered SC
  Arms: Alendronate

SUMMARY:
The main purpose of this study is to evaluate the effects of teriparatide with those of alendronate on spine bone mineral density (BMD) and other osteoporosis factors in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with osteoporosis.
* Ambulatory, 5 years or more past menopause.
* BMD T score between -2.5 and -4.0 at the lumbar spine or femoral neck.
* Normal or clinically insignificant abnormal laboratory values, including serum calcium, parathyroid hormone (PTH) 1-84, 25-hydroxyvitamin D, and alkaline phosphatase.

Exclusion Criteria:

* Prior treatment with PTH or a PTH analogue.
* Treatment with bisphosphonates within 12 months, anabolic corticosteroids or calcitriol or vitamin D analogues or agonists within 6 months, estrogens or selective estrogen receptor modulators within 3 months, or calcitonin within 2 months; therapeutic doses of fluoride; systemic corticosteroid use within 1 month or for more than 30 days in the prior year; use of anticoagulants within 1 month.
* History of diseases other than postmenopausal osteoporosis that affect bone metabolism.
* History of an increased risk of osteosarcoma (ie, patients with Paget disease of bone, previous skeletal exposure to external beam radiotherapy, or previous malignant neoplasm involving the skeleton).
* Malignant neoplasms within 5 years; carcinoma in situ of the uterine cervix within 1 year.
* Nephrolithiasis or urolithiasis within 2 years, or impaired renal function.
* Abnormal uncorrected thyroid function.
* Liver disease or clinical jaundice.
* Alcohol or other drug abuse.
* Poor medical or psychiatric risk for treatment.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2001-04; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline to 18 Months in Lumbar Spine BMD | Baseline, 18 Months

SECONDARY OUTCOMES:
Percent Change from Baseline in Lumbar Spine BMD | Baseline, 3 Months, 6 Months, 12 Months
Percent Change from Baseline in Total Hip and Femoral Neck BMD | Baseline, 12 Months, 18 Months
Percent Change from Baseline in Trabecular Volumetric BMD at the Lumbar Spine | Baseline, 6 Months, 18 Months
Percent Change from Baseline in Cortical BMD at the Femoral Neck | Baseline, 6 Months, 18 Months
Percent Change from Baseline in Trabecular BMD at the Femoral Neck | Baseline, 6 Months, 18 Months
Percent Change from Baseline in Biochemical Marker -Serum Procollagen I C-Terminal Propeptide (PICP) | Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Percent Change from Baseline in Biochemical Marker -Serum Procollagen I N-Terminal Propeptide (PINP) | Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Percent Change from Baseline in Biochemical Marker -Bone-Specific Alkaline Phosphatase (BSAP) | Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Percent Change from Baseline in Biochemical Marker -Urinary N-Telopeptide (NTX) | Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Percentage of Participants with Nonvertebral Fractures | 18 Months
Percentage of Participants with Clinical Fractures | 18 Months
Change from Baseline on the Back Pain Questionnaire | Baseline, 3 Months, 6 Months, 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Boylston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arden Hills, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morristown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providence, Rhode Island
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Recife
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mezzanine
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico